CLINICAL TRIAL: NCT01380041
Title: Identification of Multiple Sclerosis Biomarkers in Human CSF by Means of Cytokine Array
Brief Title: Cytokine in Cerebrospinal Fluid (CSF) From Multiple Sclerosis Patients
Acronym: CYTOSEP
Status: Terminated | Type: Observational
Why Stopped: Results obtained are sufficient for a publication.
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 8669; 2010-AO1321-38 (Other: Number ID-RCB)
Record Dates: First submitted 2011-06-17; First posted 2011-06-27 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2011-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosisCerebrospinal fluidBiomarkerCytokineArray
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
Multiple Sclerosis (MS) is an inflammatory disease of the brain leading to disability. Brain MRI is very useful for MS diagnosis but prognostic biomarkers are still needed. New therapies are also expected to improve MS care. Cytokine arrays provide measure of many different inflammation-related molecules that could help understanding the disease. Moreover, individual prognosis could be linked with the level of such molecules in the CSF of MS patients. The investigators will analyze the cytokine profile of MS and control patients CSF to determine a specific profile of MS and look for prognosis implication in a cohort of patients with clinically isolated syndromes (first manifesatation of MS).

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is an inflammatory disease of the brain leading to disability. Early treatment could allow better prognosis for the patients in the long term by reducing relapses rates and neurological palsy. However, individual prognostic biomarkers are still needed to adapt the treatment to a given patient. CSF is a strategic body fluid to explore in neurological diseases. In MS, it contains an elevated IgG index and/or oligoclonal bands reflecting the intrathecal synthesis of Igs around the brain. The levels of other inflammatory molecules such cytokines and metalloproteases are also known to be elevated in MS (GM-CSF, IL-6, IL-10, MMP-2, MMP9, TIMP-1, TNF-α, RANTES, MCP-1 and MIP-1). These molecules can now be easily measured by protein arrays.The aim of this study is to measure the level of 40 cytokines and 10 MMPs by means of protein arrays in the CSF from clinically definite MS (CDMS) patients, control patients and patients with a clinically isolated syndrome (CIS). The best MS markers will be determined using multiple ROC curves. Markers of rapid conversion to CDMS after a CIS will also be looked for.The best MS candidate biomarkers will be analyzed by ELISA in a new cohort of patients being recruited.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite Multiple sclerosis patients (at least 2 relapses)
* Patient having presented another neurological episode suggestive of MULTIPLE SCLEROSIS confirmed or not by a neurologist and allowing to establish the diagnosis of MULTIPLE SCLEROSIS according to the criteria of Mc Donald
* Age ≥ 18 years
* Patients informed about the objectives of the study and about its practical realization

Exclusion Criteria:

* Patient having received a treatment by corticoids in 30 days before the lumbar puncture
* Contraindication of the lumbar puncture such as an anticoagulating oral treatment for example
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically definite Multiple sclerosis patients (at least 2 relapses)Control patients (lumbar puncture for headache…
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2011-06; Primary Completion 2011-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Identification of SEP markers | 24 months
  The aim of this study is to measure the level of 40 cytokines and 10 MMPs by means of protein arrays in the CSF from clinically definite MS (CDMS) patients, control patients and patients with a clinically isolated syndrome (CIS). The best MS markers will be determined using multiple ROC curves.

CONTACTS AND LOCATIONS:
Overall Officials: Eric THOUVENOT, MD-PhD, Principal Investigator — CHRU Montpellier
Locations (1):
- CHU Montpellier, Montpellier, France